CLINICAL TRIAL: NCT05115760
Title: Intervention With Pea Protein Oral Nutrition Supplement Meal Replacement to Reduce Therapeutic Gastrostomy Tube Rates in Patients With Head and Neck Cancer Undergoing Chemoradiation Therapy
Brief Title: Pea Protein Oral Nutrition Supplement for the Reduction of Gastrostomy Tube Placement Rate in Patients With Locally Advanced Head and Neck Cancer Undergoing Chemoradiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Kate Farms Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-002182; NCI-2021-03612 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-05-14; First posted 2021-11-10 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Head and Neck Carcinoma
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive care (pea protein oral nutrition supplement) (Experimental): Patients receive Kate Farms pea protein oral nutrition supplement PO during their mealtimes as directed by their clinical dietitian during and up to 1 month following chemoradiation in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: Dietary Supplement; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Given Kate Farms pea protein oral nutrition supplement PO
  Other Names: Dietary Supplements; Nutritional Supplement; Supplement; supplemental nutrition; Supplements
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of a plant-based oral nutrition supplement, Kate Farms Standard 1.4 and/or Standard 1.0. as a primary source of nutrition in reducing the gastrostomy tube placement rate in patients with head and neck cancer that has spread to nearby tissue or lymph nodes (locally advanced) and who are undergoing chemoradiation therapy. Gastrostomy tube (G-tube) placement can be used for enteral feedings and may lead to long term side effects such as swallowing dysfunction and lead to higher rates of permanent G-tube dependence. The Kate Farms pea protein oral nutrition supplement is formulated with organic, planted-based protein for easier digestibility without artificial sweeteners or additives and without common allergens such as dairy, soy, gluten or corn. It is nutritionally complete, calorie and protein dense and available in multiple flavors that can be consumed directly or as a base for other recipes. Giving pea protein oral nutrition supplement may provide nutritional support to decrease the need for therapeutic G-tube rate during chemoradiation compared to standard supportive care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the therapeutic G-tube placement rate during chemoradiation.

SECONDARY OBJECTIVES:

I. To determine percent weight change during and following treatment. II. To determine body mass index (BMI) changes during and following treatment. III. To determine changes in nutrition status based on Global Leadership Initiative on Malnutrition (GLIM) criteria IV. To determine lean body mass before and after treatment via psoas muscle surrogate measurement on routine staging scans.

V. To determine the adherence rate of Kate Farms oral nutritional replacement. VI. To determine changes in oral and gastrointestinal microbiota via 16s ribosomal ribonucleic acid (RNA) sequencing during and following treatment in an exploratory analysis.

VII. To determine changes in biomarkers during treatment. VIIa. Serum human papillomavirus (HPV) deoxyribonucleic (DNA). VIIb. 38-multiplex immune cytokine and chemokine panel in an exploratory analysis.

VIIc. Complete metabolic panel, complete blood count with differential, C-reactive protein (CRP).

VIId. Radiosensitivity germ-line biomarker panel. VIII. To determine physician-reported acute and late toxicities during and following treatment.

VIIIa. Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. IX. To determine patient-reported quality of life during and following treatment.

IXa. University of Washington and Functional Assessment of Cancer Therapy questionnaires.

IXb. Functional Assessment of Cancer Therapy-Head & Neck (FACT-H&N). X. To determine clinical outcomes from treatment. Xa. Local/Locoregional control. Xb. Distant metastasis-free survival. Xc. Overall survival.

OUTLINE:

Patients receive Kate Farms pea protein oral nutrition supplement orally (PO) during their mealtimes as directed by their clinical dietitian during and up to 1 month following chemoradiation in the absence of unacceptable toxicity.

After completion of study intervention, patients are followed up for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented locally advanced head and neck malignancies for which concurrent chemoradiation has been recommended for definitive or adjuvant treatment
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) <= 2
* Body mass index > 18kg/m^2
* No evidence of distant metastatic disease (M1 disease)
* No G-tube placement prior to initiation of chemoradiation
* Eligible to undergo concurrent chemotherapy as determined by treating oncologist
* If a woman is of childbearing potential, a negative urine pregnancy test must be documented prior to proceeding with chemoradiation. Women of childbearing potential must agree to use medically acceptable forms of adequate contraception (hormonal or barrier method of birth control; or abstinence) for the entire study period and for up to 4 weeks after study treatment
* While negative pregnancy would be verified by urine test routinely prior to chemo-radiation therapy, we do not ask for verification of a negative urine pregnancy test.
* Ability to understand and willingness to sign a written informed consent
* Able to tolerate the taste of the Kate Farms Standard 1.4 or Standard 1.0 oral nutritional supplement at the time of screening
* Able and willing to participate in the Swallow Preservation Program at the Speech Pathology Clinic
* No evidence of clinically significant swallowing dysfunction by history or physical exam at time of radiation oncology consultation

Exclusion Criteria:

* Patients who refuse to use Kate Farms oral nutritional meal replacement due to its taste or other patient preference reasons
* Patients with allergies to any of the ingredients contained in Kate Farms nutritional replacement
* Evidence of clinically significant swallowing dysfunction by history or physical exam at time of radiation oncology consultation
* Refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Compliance rate | Up to 1 month post chemoradiation
  Will calculate the compliance rate and the corresponding 95% exact confidence interval.
Gastrostomy (G)-tube placement rate | Up to 1 month post chemoradiation
  Will calculate the compliance rate and the corresponding 95% exact confidence interval. The 95% exact confidence interval (CI) will be provided.

SECONDARY OUTCOMES:
Weight change measurement | Up to 2 years
  Weight data will be collected at each visit and summary descriptive statistics will be calculated at each time points. Repeated measure analysis of variance (ANOVA) will be used to explore if there are any change in these parameters over time. Treatment breaks will be recorded in days per study patient and summarized. G-tube placement timing will be recorded for patients receiving G-tubes, and the duration of G-tube dependence will be recorded in days per study patient and summarized.
Body mass index change measurement (BMI) | Up to 2 years
  BMI data will be collected at each visit and summary descriptive statistics will be calculated at each time points. Repeated measure ANOVA will be used to explore if there are any change in these parameters over time. Treatment breaks will be recorded in days per study patient and summarized. G-tube placement timing will be recorded for patients receiving G-tubes, and the duration of G-tube dependence will be recorded in days per study patient and summarized.
Global Leadership Initiative on Malnutrition criteria | Up to 2 years
  Will be collected at each visit and summary descriptive statistics will be calculated at each time points. Repeated measure ANOVA will be used to explore if there are any change in these parameters over time. Treatment breaks will be recorded in days per study patient and summarized. G-tube placement timing will be recorded for patients receiving G-tubes, and the duration of G-tube dependence will be recorded in days per study patient and summarized.
Patient-reported quality of life (QOL): The University of Washington Quality of Life Questionnaire (UW-QOL). | Up to 2 years
  Patient-reported QOL according to the University of Washington (UW-QOL) questionnaires will be summarized by descriptive statistics by visit time points.
  The University of Washington Quality of Life Questionnaire (UW-QOL) is a self-administered scale measuring health-related quality life specifically for head and neck cancer patients. It is scored from 0-100 with higher scores indicating a better quality of life.
Patient-reported quality of life (QOL): The Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN). | Up to 2 years
  Patient-reported QOL according to the Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) questionnaires will be summarized by descriptive statistics by visit time points.
  Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) is a 12 item self-administered scale measuring health-related quality of life specifically for head and neck cancer patients. Response options form a Likert scale and a subscale score is computed by summing across all items, with higher scores reflecting better QOL.
Local/locoregional control | Up to 2 years
  Will be estimated using the Kaplan-Meier method.
Distant metastasis-free survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method.
Overall survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method.
Incidence of adverse events (AEs) | Up to 2 years
  Toxicity will be graded using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version (v) 4.0. AEs and serious (S)AEs will be reported using a CTCAE v 4.0 terminology and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States